CLINICAL TRIAL: NCT00309075
Title: Multicenter, Open-label Study of the Safety (Open-label) and Efficacy (Open-label and Blinded Reader) of a Single Administration of Approximately 0.1 mmol/kg of Magnevist® Injection-enhanced Magnetic Resonance Arteriography (MRA) and 2-dimensional-time-of-flight (2D-TOF) MRA in Patients With Known or Suspected Disease of the Calf and/or Pedal Arteries Undergoing MRA of the Calf and Pedal Arteries With Intra-arterial Digital Subtraction Arteriography (i.a. DSA) as the Standard of Reference.
Brief Title: Magnevist® Injection Enhanced MRA Compared to Non Contrast MRA for the Detection of Stenosis in the Calf and/or Pedal Arteries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 91251; 307260
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Stenosis
Keywords: Stenosis of the calf and/or pedal arteries
MeSH Terms: conditions — Constriction, Pathologic | interventions — Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Gadopentetate dimeglumine (Magnevist)

INTERVENTIONS:
Drug: Gadopentetate dimeglumine (Magnevist) — Gadopentetate dimeglumine (Magnevist Injection), approximately 0.1mmol/kg body weight, single intravenous administration on the study day

SUMMARY:
The purpose of this study is to look at the safety (what are the side effects) and efficacy (how well does it work) of Magnevist (the study drug) used for MRI of the calf and foot arteries. The results will be compared to the results of MRI taken without Magnevist, and with the results of your X-ray angiography.

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.Bayer HealthCare Pharmaceuticals, Inc.is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Has known or suspected disease of the calf and/or pedal arteries
* Is scheduled for X-ray angiography

Exclusion Criteria:

* Has any contraindication to magnetic resonance imaging
* Is scheduled for any procedure before the X-ray angiography
* Had previously had stents placed bilaterally in the calf and/or foot arteries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2003-12; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Accuracy, sensitivity, and specificity based on visual assessment of stenosis assesses by blinded reader | Image creation after injection - evaluation at blind read

SECONDARY OUTCOMES:
Diagnostic confidence | At blinded and/or open label read of the images
Accuracy, sensitivity, and specificity based on visual assessment of stenosis assesses by open label reader | At blinded and/or open label read of the images
Location and matching of stenosis | At blinded and/or open label read of the images
Image quality | At blinded and/or open label read of the images
Image evaluability and presence of artefacts | At blinded and/or open label read of the images
Ability to visualize arteries | At blinded and/or open label read of the images
Exact categorization of stenosis | At blinded and/or open label read of the images
Number of evaluable arteries | At blinded and/or open label read of the images
Duration of 2D-TOF and MRA | At blinded and/or open label read of the images
Artery appropriate for bypass | At blinded and/or open label read of the images
Patient management | from baseline to 24 hours follow-up
Safety | from baseline to 24 hours follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer